CLINICAL TRIAL: NCT04755907
Title: Validation of the Three-dimensional Bioprinted Tumor Models as a Predictive Method of the Response to Chemotherapy for Colorectal Cancer With or Without Liver Metastases
Brief Title: 3D Bioprinted Models for Predicting Chemotherapy Response in Colorectal Cancer With/Without Liver Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRC-3D-Bioprint
Record Dates: First submitted 2021-02-13; First posted 2021-02-16 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Colorectal Cancer Liver Metastasis
Keywords: colorectal cancer; colorectal cancer liver metastasis; three-dimensional bioprinting; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — resected tumor tissue from surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: colorectal cancer patients at resectable stage II/III who will receive adjuvant chemotherapy after surgery
  Interventions: Procedure: surgical resection; Other: adjuvant chemotherapy
- Group B: colorectal cancer patients at locally advanced stage who will receive neoadjuvant chemotherapy before surgery and adjuvant chemotherapy after surgery
  Interventions: Procedure: surgical resection; Other: adjuvant chemotherapy; Other: neoadjuvant therapy
- Group C: colorectal cancer patients with liver metastases
  Interventions: Procedure: surgical resection; Other: adjuvant chemotherapy; Other: neoadjuvant therapy

INTERVENTIONS:
Procedure: surgical resection — Surgical resection will be performed for locoregional lesions or liver metastases.
Other: adjuvant chemotherapy — Regimens of adjuvant chemotherapy are directed by clinical guidance and experience.
Other: neoadjuvant therapy — Regimens of neoadjuvant chemotherapy are directed by clinical guidance and experience.
  Groups: Group B; Group C

SUMMARY:
The therapeutic regimens of adjuvant and neoadjuvant chemotherapy for colorectal cancer (CRC) remain largely relied on clinical experience, and thus preclinical models are needed to guide individualized medicine. The investigators are going to establish 3D bioprinted CRC models and organoids from surgically resected tumor tissues of CRC patients with or without liver metastases. In vitro 3D models and organoids will be treated with the same chemotherapy drugs with the corresponding patients from whom the models are derived. The sensitivity of chemotherapy drugs will be tested in these two types of in vitro models, and the actual response to chemotherapy in patients will be evaluated. The predictive ability of 3D models for chemotherapy sensitivity in CRC patients will be compared with that of the organoids. This observational study will validate the potential value of 3D bioprinted tumor models in predicting the response to chemotherapy in CRC.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Diagnosed as colorectal cancer with or without liver metastases before
* Pathologically proven colorectal cancer after surgery

Exclusion Criteria:

* Medical history with other malignancies or serious diseases
* Disable to sign the informed consent independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically and pathologically proven colorectal cancer patients are considered as potential candidates of this study. Medical history will be thouroughly taken by clincal practicitioners. Only patients older than 18 years will be included. Those with medical hostory of other malignancies or serious diseases will be excluded. Patients who are not able to sign the informed consent independently will not be included in this study. All the patients included in this study will receive adjuvant/neoadjuvant chemotherapy and surgical resection for the treatment of CRC.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response of 3D tumor models/organoids to the same chemotherapy drugs as the corresponding patients. | 2021.03-2021.12
  The investigators will establish and culture 3D colorectal cancer models and organoids. The 3D models and organoids will be treated with the same chemotherapy drugs as the corresponding patients. The viability of the 3D tumor models and organoids will be observed after treatment and the IC50 of each drug will be calculated. The correlation of 3D model/organoid sensitivity and the patient response will be analyzed.

SECONDARY OUTCOMES:
Response of the colorectal cancer patients to neoadjuvant chemotherapy. | 2021.03-2022.03
  For patients who receive neoadjuvant chemotherapy before surgery, the response to neoadjuvant chemotherapy will be evaluated according to clinical imaging results and the RECIST scores.

OTHER OUTCOMES:
Response of the colorectal cancer patients to adjuvant chemotherapy. | 2021.03-2023.12
  The response to adjuvant chemotherapy will be evaluated according to disease free survival (DFS). Regular follow-ups will be conducted, and DFS is difined as the interval between the date of surgery and the date of last follow-up or recurrence/progression.

CONTACTS AND LOCATIONS:
Overall Officials: Yilei Mao, MD PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) can be accessed with reasonable requests via e-mail. IPD will be shared after the study is completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will available after the study is completed.
Access Criteria: Data can be accessed via e-mail with reasonable requests.

REFERENCES:
- [Background] Wu J, Lu AD, Zhang LP, Zuo YX, Jia YP. [Study of clinical outcome and prognosis in pediatric core binding factor-acute myeloid leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2019 Jan 14;40(1):52-57. doi: 10.3760/cma.j.issn.0253-2727.2019.01.010. Chinese. PMID 30704229
- [Background] Brancato V, Oliveira JM, Correlo VM, Reis RL, Kundu SC. Could 3D models of cancer enhance drug screening? Biomaterials. 2020 Feb;232:119744. doi: 10.1016/j.biomaterials.2019.119744. Epub 2019 Dec 26. PMID 31918229
- [Background] Bruun J, Kryeziu K, Eide PW, Moosavi SH, Eilertsen IA, Langerud J, Rosok B, Totland MZ, Brunsell TH, Pellinen T, Saarela J, Bergsland CH, Palmer HG, Brudvik KW, Guren T, Dienstmann R, Guren MG, Nesbakken A, Bjornbeth BA, Sveen A, Lothe RA. Patient-Derived Organoids from Multiple Colorectal Cancer Liver Metastases Reveal Moderate Intra-patient Pharmacotranscriptomic Heterogeneity. Clin Cancer Res. 2020 Aug 1;26(15):4107-4119. doi: 10.1158/1078-0432.CCR-19-3637. Epub 2020 Apr 16. PMID 32299813
- [Background] Yao Y, Xu X, Yang L, Zhu J, Wan J, Shen L, Xia F, Fu G, Deng Y, Pan M, Guo Q, Gao X, Li Y, Rao X, Zhou Y, Liang L, Wang Y, Zhang J, Zhang H, Li G, Zhang L, Peng J, Cai S, Hu C, Gao J, Clevers H, Zhang Z, Hua G. Patient-Derived Organoids Predict Chemoradiation Responses of Locally Advanced Rectal Cancer. Cell Stem Cell. 2020 Jan 2;26(1):17-26.e6. doi: 10.1016/j.stem.2019.10.010. Epub 2019 Nov 21. PMID 31761724
- [Background] Xie F, Sun L, Pang Y, Xu G, Jin B, Xu H, Lu X, Xu Y, Du S, Wang Y, Feng S, Sang X, Zhong S, Wang X, Sun W, Zhao H, Zhang H, Yang H, Huang P, Mao Y. Three-dimensional bio-printing of primary human hepatocellular carcinoma for personalized medicine. Biomaterials. 2021 Jan;265:120416. doi: 10.1016/j.biomaterials.2020.120416. Epub 2020 Sep 22. PMID 33007612
- [Background] Sun L, Yang H, Wang Y, Zhang X, Jin B, Xie F, Jin Y, Pang Y, Zhao H, Lu X, Sang X, Zhang H, Lin F, Sun W, Huang P, Mao Y. Application of a 3D Bioprinted Hepatocellular Carcinoma Cell Model in Antitumor Drug Research. Front Oncol. 2020 Jun 3;10:878. doi: 10.3389/fonc.2020.00878. eCollection 2020. PMID 32582546